CLINICAL TRIAL: NCT06398210
Title: Investigation of the Effectiveness of Cognitive Exercise Therapy Approach in Patients With Primary Sjögren's Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Nazli Elif Nacar, Physioterapist-MSc, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KahramanmarasSIU.
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-07

CONDITIONS: Primer Sjogren's Syndrome
Keywords: Sjogren' Syndrome; biopsychosocial model; health-related quality of life; patient-reported outcome measure; psychosocial intervention
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Intervention Model Description: Single Blinded-Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group exercise (Experimental): Patients will be included in group exercise, 36 sessions in total; He/she will attend BETY-group sessions lasting 1 hour, 3 times a week for 12 weeks.
  Interventions: Other: Cognitive Exercise Therapy Approach (BETY)
- Individual exercise (Experimental): Patients will be included in individual exercise, 36 sessions in total; He/she will attend BETY-individual sessions lasting 1 hour, 3 times a week for 12 weeks.
  Interventions: Other: Cognitive Exercise Therapy Approach (BETY)
- Control (No Intervention): In the control group, exercise recommendations will be given as a home program according to the symptoms of the individuals.

INTERVENTIONS:
Other: Cognitive Exercise Therapy Approach (BETY) — Cognitive Exercise Therapy Approach (BETY) BETY includes mind-body interaction information management, pain management strategies, mood information management through dance therapy/authentic movement, and sexuality information management. BETY first session; After meeting the patient and completing the evaluations, it consists of the steps of analysis of the person's problem, selection of exercise for this problem, replacement of the exercise in function, pain management, and recovery agreement. The basic exercise model used in BETY is function-oriented trunk stabilization exercises. Patients are given information about the 5 features of trunk stabilization (neck, shoulder, rib cage, lumbopelvic region postures, and respiratory control), visual imagery, and their control.
  Arms: Group exercise; Individual exercise

SUMMARY:
To determine the effectiveness of the Cognitive Exercise Therapy Approach (BETY in Turkish) in individuals with Primary Sjögren's Syndrome and to compare the effects of this training when applied in groups and individually.

H1: BETY training affects at least one of the following: disease activity, pain, and fatigue in individuals with Primary Sjögren's Syndrome.

H2: BETY training affects at least one of the quality of life and biopsychosocial status in individuals with Primary Sjögren's Syndrome.

H3: BETY training affects the anxiety/depression level in individuals with Primary Sjögren's Syndrome.

H4: BETY training affects chewing and swallowing performances in individuals with Primary Sjögren's Syndrome.

H5: BETY training given in groups is more effective than individual practice in individuals with Primary Sjögren's Syndrome.

Volunteers who meet the inclusion criteria will be placed on the waiting list, the content of all three interventions will be explained to the individuals, and groups will be formed randomly using the sealed envelope method among those who volunteer to participate in all three contents. The three options that will be offered to patients will be 'participation in BETY group sessions', 'participation in individual BETY sessions', and 'following a home program with symptom-oriented exercise recommendations'.

The biopsychosocial-based exercise model ("Cognitive Exercise Therapy Approach" (BETY)) to be used in this randomized controlled study is a method developed on individuals with rheumatic diseases. In this method, which can be applied individually or in a group, nociplastic pain, and mood management are combined with exercises. Patients participating in the training received 36 sessions in total; He/she will attend BETY sessions lasting 1 hour, 3 times a week for 12 weeks, in group and individual sessions. Each session will include a warm-up phase, exercise training, and cool-down phases. During these sessions, the physiotherapist plays only an instructive and guiding role. In BETY sessions, exercises will be made more difficult as the person can perform a higher level exercise, in accordance with the loading principle. An exercise band will be added to the exercises that show a progression from closed kinetic chain to open kinetics, following the developments in the patient.

In the control group, exercise recommendations will be given as a home program according to the individuals' symptoms.

Cognitive Exercise Therapy Approach (BETY) BETY includes mind-body interaction information management, pain management strategies, mood information management through dance therapy/authentic movement, and sexuality information management. BETY first session; After meeting the patient and completing the evaluations, it consists of the steps of analysis of the person's problem, selection of exercise for this problem, replacement of the exercise in function, pain management, and recovery agreement. The basic exercise model used in BETY is function-oriented trunk stabilization exercises. Patients are given information about the 5 features of trunk stabilization (neck, shoulder, rib cage, lumbopelvic region postures and respiratory control), visual imagery, and their control.

BETY-nociplastic pain management strategy includes the following steps;

* Physical activity is stopped when there is pain.
* Due to the relationship between pain and central sensitization, the patient questions whether he or she is worried about something. If there is a situation that causes concern, the patient should direct his/her attention away from this point.
* Cognitive restructuring is achieved with positive thoughts instead of negative thoughts as a distraction strategy.
* At the moment of positive thought, it is recommended to do exercises for the painful area.

Information management in sexuality means that anxiety about sexuality is also a factor that increases pain.

It is added to the sessions with the knowledge that it may be a factor and because it is a subject that cannot usually be talked about. During the "arm openings 1" and "arm openings 2" exercises, during the cognitive restructuring process using positive and negative awareness sentences, is aimed at normalizing these issues in the mind of the individual by including positive and negative sentences about sexuality. In addition, the information will be reinforced by synthesizing the questions asked by the patients during patient education and the pelvic floor muscle training created by trunk stabilization exercises.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Primary Sjögren's Syndrome
* 18 years or older

Exclusion Criteria:

* Patients with Secondary Sjögren's Syndrome,
* Participated in a regular exercise program in the last 2 months,
* Patients who are diagnosed with other uncontrolled/clinically important diseases (chronic obstructive pulmonary disease, congestive heart failure, endocrine system diseases, neurological, psychological diseases, etc.),
* Having a malignant condition,
* Pregnant individuals,
* Have other conditions that prevent exercise,
* Individuals who do not agree to participate in the study and do not give written consent will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
BETY-Biopsychosocial Questionnaire (BETY-BQ) | baseline-12. week-6. month
  BETY-BQ consists of the following six subtitles that investigate in detail the biopsychosocial dimensions: pain, functionality and fatigue, mood, sociability, sexuality, and sleep quality. This scale consists of 30 items, scored on a 5-point Likert system. Each question is scored as "No never: 0 Yes rarely: 1 Yes sometimes: 2 Yes often: 3 Yes always: 4" and a total score over 30 items. A higher score indicates a poorer biopsychosocial situation.

SECONDARY OUTCOMES:
Central Sensitization Scale | baseline-12. week-6. month
  In this scale, which consists of 40 questions and questions the symptoms related to central sensitization, a score above 40 is interpreted as an indicator of central sensitization. Turkish validity and reliability study was conducted.
Pain Catastrophizing Scale | baseline-12. week-6. month
  It is a Likert-type self-assessment scale consisting of 13 items. Each item is scored between 0 and 4 points. The total score ranges from 0 to 52. High scores indicate a high level of catastrophizing. It has 3 subtests: pain magnification (items 6, 7 and 13), rumination (items 8, 9, 10, 11) and helplessness (items 1, 2, 3, 4, 5 and 12). Turkish validity and reliability study was conducted.
EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) | baseline-12. week-6. month
  ESSDAI is a clinical scale that measures disease activity in Sjögren's Syndrome and its items provide objective data consisting of tests applied to patients during routine outpatient clinic check-ups. An ESSDAI score of less than 4 indicates low activity, a score between 5 and 13 indicates moderate activation, and a score of 14 and above indicates high activity.
EULAR Sjögren's Syndrome Patient Reporting Index (ESSPRI) | baseline-12. week-6. month
  ESSPRI scoring is a symptom severity assessment scale filled out by the patient and used in Sjögren's Syndrome. The patient is asked to express fatigue, pain and dryness complaints with a score between one and ten, and the arithmetic average of the score obtained from these three questions forms the result. An ESSPRI score of less than 5 is considered an acceptable disease state, while a score of 5 or above is considered a sign of high activity.
Hospital Anxiety and Depression Scale (HADS) | baseline-12. week-6. month
  In this scale consisting of fourteen questions, odd-numbered questions question anxiety, and even questions question depression. Options range from 0 to 3, with a higher score indicating a poor emotional state. The cut-off values of the scale were determined as 10 for the anxiety subscale and 7 for the depression subscale. Turkish version study was conducted.
Primary Sjögren's Syndrome Quality of Life Scale | baseline-12. week-6. month
  This scale, consisting of twenty-five questions, is divided into two subsections: physical (discomfort and dryness) and psychosocial. Since vaginal dryness, one of the symptoms of SS, was included in the total score, the maximum score was determined as 96 for women and 92 for men. A high score means low health-related quality of life.
Multidimensional Fatigue Rating Scale | baseline-12. week-6. month
  This scale evaluates fatigue with 16 items under 5 subheadings: degree, severity, impact on daily activities, troubles it causes and fatigue time. The score ranges from 0 (not tired) to 50 (extremely tired). The Turkish validity and reliability study of the scale was conducted.
Turkish Eating Assessment Tool (T-EAT-10) | baseline-12. week-6. month
  T-EAT-10 is a survey consisting of 10 questions with a Likert scale between 0 and 4 (0 = no problem, 4 = severe problem). The total score is calculated out of 40 points by finding the sum of the answers given by individuals to each question. A score of 3 or more in the survey is considered abnormal. A score of 16 or above is considered as suspicion of aspiration. Turkish validity and reliability were tested.
Yale Swallow Protocol | baseline-12. week-6. month
  Yale Swallow Protocol is a reliable screening test performed under expert supervision to determine the risk of aspiration at an early stage. The protocol has three main components. These are exclusion criteria, a short cognitive test, and oral mechanism, and drinking 3 oz (90 cc) water directly from the glass or with a straw. Risk factors are examined in the 1st and 2nd stages to determine the patients to whom the test can be applied. Patients who complete step 1 and are not contraindicated for testing proceed to the short cognitive testing phase. Patients who pass the short cognitive test and oral mechanism stages can proceed to the third stage, which is drinking 90 cc of water. The 90 cc water swallow challenge protocol is a simple assessment that can be used by many qualified healthcare professionals to identify aspiration risk because it is easy to perform, highly reliable, cost-effective, and clinically validated.Patients showing these findings are recorded as 'failing' the test.
Test of Mastication and Swallowing Solids | baseline-12. week-6. month
  In our study, the Test of Mastication and Swallowing Solids (TOMASS) will be used. The test evaluates how many bites the individual takes to eat a biscuit while sitting upright, how many chewing cycles he makes, how many times he swallows it, and how long the total time is from biting to swallowing. Video recording will be taken during the test. The number of bites, number of chewing cycles, number of swallows and total time will be calculated on the video. Individuals will be asked to eat the biscuit normally while sitting on a chair in an upright position with the throat visible. Meanwhile, video recording will be taken from the individuals' front view, showing their mouth and neck. The evaluation of the test will then be made by the evaluator. Videos will be stored in folders on an encrypted computer and only the work team will have access.
Dysphagia limit | baseline-12. week-6. month
  While evaluating dysphagia, individuals are given 5, 10, 15, 20, 25, 30, 35, 40 and 45 mL volumes of liquid, respectively, with a graduated syringe and are asked to swallow the liquid. The maximum amount of fluid that the thyroid cartilage can swallow during a single movement is determined. The normal dysphagia limit in healthy individuals is more than 20 mL. If a person can swallow 20 mL normally, the dysphagia limit is normal.
Xerostomia inventory | baseline-12. week-6. month
  The scale consists of 11 items. Patients will be asked to choose the best response for each item describing their symptoms over the previous two weeks. Responses are scored from 1 to 5 (1: never, 2: rarely, 3: occasionally, 4: fairly often, and 5: very often). The sum of the item scores gives a total score ranging from 11 to 55, and a higher score indicates that the symptoms are more severe. The Turkish validity and reliability study of the scale in individuals with primary Sjögren's Syndrome was conducted.

CONTACTS AND LOCATIONS:
Locations (1):
- Nazli Elif Nacar, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No